CLINICAL TRIAL: NCT03135977
Title: A Clincal Trial of Apatinib Mesylate and Etoposide(VP-16) as the Maintenance Therapy in Extensive-stage Small Cell Lung Cancer After First-line Chemotherapy
Brief Title: Apatinib and Etoposide as the Maintenance Therapy in Extensive-stage Small Cell Lung Cancer After First-line Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, xionghong cai, epartment of Medical Oncology, Sichuan Cancer Hospital & Institute, Chengdu, Sichuan, PR China, Sichuan Cancer Hospital and Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Ahead-SL-20170220
Record Dates: First submitted 2017-04-27; First posted 2017-05-02 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Extensive-stage Small Cell Lung Cancer; Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms | interventions — apatinib; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib, Etoposide (Experimental): Patients receive etoposide 50mg from day 1 to day 14 and apatinib 250mg/d from day 1 to day 21, repeated every 21 days until progressive Disease(PD) .
  Interventions: Drug: Apatinib, Etoposide

INTERVENTIONS:
Drug: Apatinib, Etoposide — Patients receive etoposide 50mg from day 1 to day 14 and apatinib 250mg/d from day 1 to day 21, repeated every 21 days until progressive Disease(PD) .
  Other Names: VP-16

SUMMARY:
Although fist-line therapy with Cisplatin and etoposide(EP)or Carboplatin and etoposide(CE) has been given, patients with extensive small cell lung cancer(ED-SCLC) still relapse and the 2-year survival is extremely low. There is no standard maintenance treatment recommendation for ED-SCLC patients after the first-line therapy.Apatinib has been approved as a second-line treatment for advanced gastric cancer. Several phase III clinical studies of non small cell lung cancer, liver cancer, colorectal cancer and other tumors also showed apatinib has less toxic side effects and better patient tolerance. However, the clinical application of apatinib in small cell lung cancer is still lack of evidence-based medicine,so this clinical trial is designed to investigate the efficacy and safety of apatinib combine with etoposide as maintenance therapy in ED-SCLC patients after first-line chemotherapy in our center.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of extensive-stagesmall cell lung caner(SCLC) ,after first-line therapy
* Performance status of 0～2 on the ECOG criteria
* Expected survival is above three months
* Adequate hematologic (neutrophil count>=1.5×109/L, hemoglobin>=80g/L, platelets>=80×109/L), hepatic function (aspartate transaminase (AST) & alanine transaminase(ALT) =<upper normal limit(UNL) x2, bilirubin level =< UNL x 1.5)
* Patients have the ability to understand and voluntarily sign the informed consent, and allow adequate follow-up.

Exclusion Criteria:

* suffered from other tumor within 5 years( Except: cervical carcinoma in situ, cured basal cell carcinoma, cured bladder epithelial tumor).
* Difficulties in taking pills (inability to swallow tablets,GI tract resection, chronic bacillary diarrhea and intestinal obstruction).
* Bleeding tendency or coagulation disorders.
* Uncontrolled hypertension (systolic pressure>150 mmHg , or diastolic pressure> 90 mmHg).
* Urine protein≥++, or urine protein in 24 hours≥2.0g.
* severe uncured wounds, ulcers or fracture.
* Pregnant or breast-feeding.
* Patients with epilepsy who need to take medicine (such as steroids or anti epilepsy agents).
* The researcher believe that the Patient is not suitable to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 6 months
  The first day of treatment to the date that disease progression is reported

SECONDARY OUTCOMES:
Overall survival | up to 24 months
  the first day of treatment to death or last survival confirm date
Duration of Response | up to 24 months
  Duration of response is defined as time from the date of the first observed hematologic improvement to the date of the first subsequent documented disease progression or relapse
Tumor response rate | Time Frame: 3 month
  The ratio between the number of responders and number of patients assessable for tumor response.
Quality of Life (QoL) questionnaire | up to 24 months
  in cancer patients and survivors with dermatologic conditions. This is a nontherapeutic and nondiagnostic protocol to obtain quality of life assessments from cancer patients and survivors who have dermatologic conditions, whether related to cancer therapies, or directly related to the primary cancer diagnosis. Data will be collected by using one or more dermatology-specific QoL instruments based on the underlying skin condition/s.

CONTACTS AND LOCATIONS:
Overall Officials: Xionghong Cai, Doctor, Principal Investigator — Sichuan Cancer Hospital and Research Institute
Locations (1):
- Sicchuan cancer hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided